CLINICAL TRIAL: NCT01839565
Title: A Prospective and Retrospective Multicenter Registry for Surgeon-based Evaluation of the "Quadrilateral Surface Plate" Used for Acetabular Fractures
Brief Title: Quadrilateral Surface Plate (QSP) Focused Registry
Status: Completed | Type: Observational
Sponsor: AO Clinical Investigation and Publishing Documentation (Other)
Responsible Party: Sponsor
Organization: AO Innovation Translation Center (Other)
Other Study IDs: FR_QSP
Record Dates: First submitted 2013-04-12; First posted 2013-04-25 (Estimated); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Acetabular Fracture
Keywords: Adverse events; Osteosynthesis; Quality of life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients undergoing osteosynthesis of acetabular fractures by using the Quadrilateral Surface Plate
  Interventions: Device: Quadrilateral Surface Plate

INTERVENTIONS:
Device: Quadrilateral Surface Plate — Patients with acetabular fracture surgically treated using the Quadrilateral Surface Plate

SUMMARY:
The absence of methodologically, prospectively and retrospectively collected information on the use of the Quadrilateral Surface Plate (QSP) in the given indication requires a multicenter approach. Using a registry to get more information about the effectiveness and possible benefits or complications during the surgery and during the post-operative treatment is adequate and necessary to get new insights to the use of the Quadrilateral Surface Plate.

DETAILED DESCRIPTION:
This registry includes six visits at which data is collected form the patinet (pre-op, post-op, 6 weeks FU, 3 months FU, 6 months FU and 12 months FU). Patients can be inlucded prospectively or retrospectively. If properatively recruited patients complete two questionnaires (EQ5D and Merle d'Aubigné) at their preoperative visits. These questionnaires are repeated after 6 and 12 months. Surgeons report about the success of the surgical procedure in a specifically designed questionnaire.

During the whole study period, adverse events related to the implant or surgery are collected as well as x-rays and CT (as per standard of care).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of acetabular fracture requiring surgical fixation
* Ability to understand the content of the patient information / informed consent form
* Signed and dated IRB/EC-approved written informed consent

Exclusion Criteria:

* Any not medically managed severe systemic disease
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Prisoner
* Participation in any other medical device or medicinal product registry within the previous month that could influence the results of the present registry

Intraoperative exclusion criteria:

* Intraoperative decision to use implants other than the device under investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The increasing number of acetabular fractures in elderly individuals with osteoporosis has added new technical challenges to surgical management. A common group of fracture patterns in this population is the anterior wall or column often with an associated posterior hemitransverse.
  These injuries frequently also include quadrilateral surface comminution which can make both reduction and stabilization more difficult. The 3.5 mm quadrilateral surface plate was developed to provide a more effective way to deal with these issues, for example, a way to deal with the quadrilateral surface enbloc for reduction, allowing buttress stabilization, which is independent of bone density.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-10; Primary Completion 2017-03 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Surgical treatment-related Adverse Events | Intra-operative
  Collection of (Serious) Adverse Events related to the surgical treatment of the acetabular fracture.

SECONDARY OUTCOMES:
Changes in Quality of Life | Post-op till Hospital Discharge; 6 weeks; 3, 6, 12 and 24 months post-operative
  Changes in Quality of Life, pain and mobility using questionnaires (EQ-5D and Merle d'Aubigné score)
Fracture Healing | Post-op till Hospital Discharge; 6 weeks; 3, 6, 12 and 24 months post-operative
  Fracture healing: defined as a fracture radiographically showing at least three cortices with signs of callus or trabeculae crossing from one side of the fracture to the other.
Surgical treatment-related Adverse Events till discharge | post-operative
  Collection of surgery-related (Serious) Adverse Events related to surgical procedure at timepoint:
  - 1-12 days postoperative (till discharge)
Surgical treatment-related Adverse Events till 6 weeks | post-operative
  Collection of surgery-related (Serious) Adverse Events related to surgical procedure at timepoint:
  - 6 weeks postoperative
Surgical treatment-related Adverse Events till 3 months | post-operative
  Collection of surgery-related (Serious) Adverse Events related to surgical procedure at timepoint:
  - 3 months postoperative
Surgical treatment-related Adverse Events till 6 months | post-operative
  Collection of surgery-related (Serious) Adverse Events related to surgical procedure at timepoint:
  - 6 months postoperative
Surgical treatment-related Adverse Events till 12 months | post-operative
  Collection of surgery-related (Serious) Adverse Events related to surgical procedure at timepoint:
  - 12 months postoperative
Surgical treatment-related Adverse Events till 24 months | post-operative
  Collection of surgery-related (Serious) Adverse Events related to surgical procedure at timepoint:
  - 24 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Tim Pohlemann, Prof. MD, Principal Investigator — AO foundation
Locations (6):
- Germany (4):
  - Berufsgenossenschaftliche Unfallklinik Frankfurt am Main, Frankfurt
  - Universitaetsklinikum Heidelberg, Heidelberg
  - University of Saarland, Homburg/Saar
  - Klinikum der Johannes Gutenberg Universitaet Mainz, Mainz
- Ortopedia e Traumatologia, Rome, Italy
- Luzerner Kantonsspital, Lucerne, Switzerland